CLINICAL TRIAL: NCT00186745
Title: Tinzaparin for Treatment of Venous Thromboembolism in Renal Insufficiency: A Pilot Study
Brief Title: Use of Low Molecular Weight Heparin (Tinzaparin) to Treat Blood Clots in Patients With Kidney Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ceased
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); LEO Pharma (Industry)
Responsible Party: Principal Investigator, Wendy Lim, Associate Professor, Department of Medicine, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA 5723
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Venous Thrombosis; Pulmonary Embolism
Keywords: Venous thrombosis; Pulmonary embolism; Kidney failure; Anticoagulants; Heparin, Low-Molecular-Weight
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Renal Insufficiency | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All patients in this cohort receive treatment with weight-adjusted, standard-dose tinzaparin for treatment of venous thromboembolism. Trough anti-Xa level measurements done on any 2 of days 3, 5 or 7 of treatment. Patients with a trough anti-Xa level > 0.5 IU/mL receive dose adjustment of the tinzaparin.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — Dose: 175 IU/kg subcutaneously once daily, up to 7 days. Dose reduction as per protocol if anti-Xa levels exceed pre-defined limits.
  Other Names: Brand name: Innohep

SUMMARY:
Blood clots in the leg veins, known as deep vein thrombosis, are important because they may travel to the lung (known as pulmonary embolism) and cause death. Blood clots are treated with blood thinners, or anticoagulants. The preferred treatment is an anticoagulant known as low molecular weight heparin (LMWH). LMWH is given by an injection under the skin, which is convenient for patients because they can self-administer this medication at home, and no blood testing is required. However, LMWH is cleared from the body through the kidneys, so patients who have kidney failure are generally not treated with LMWH because they may be at a higher risk of bleeding.

One type of LMWH, known as tinzaparin, may be less dependent on the kidneys for clearance and may not increase in patients with kidney failure. The investigators would like to use tinzaparin to treat patients who have deep vein thrombosis or pulmonary embolism, and who also have kidney failure.

The purpose of this study is to determine whether the blood thinning effects of tinzaparin build up, or accumulate, in patients with varying degrees of kidney failure compared to patients without kidney failure. The blood thinning effects will be measured using a blood test known as an anti-Xa level. Patients will be followed over the time they receive tinzaparin and those patients who are found to have potentially high levels of tinzaparin (based on the anti-Xa level) will have their tinzaparin dose adjusted. The investigators believe that the levels of tinzaparin will not accumulate to potentially dangerous levels in a significant number of patients with kidney failure.

DETAILED DESCRIPTION:
Background and rationale. Venous thromboembolism (VTE) is an important clinical problem because it is common, preventable, contributes to morbidity and mortality, and is costly. Low molecular weight heparin (LMWH) is the preferred anticoagulant for VTE treatment, but is renally excreted. Consequently, LMWH use in patients with renal insufficiency may result in accumulation of the anticoagulant effects and the potential for avoidable bleeding complications. As a result, most patients with renal insufficiency who also have VTE are unable to benefit from LMWH treatment. These patients are therefore generally treated in hospital using unfractionated heparin (UFH), since it is eliminated by extra-renal mechanisms. In addition to those patients with known renal insufficiency, many elderly patients have previously unrecognized renal insufficiency and treatment of these patients with LMWH can be associated with accumulation of the anticoagulant effect and avoidable bleeding.

Tinzaparin, relative to other LMWHs, has a higher molecular weight and greater negative charge: both biochemical features that favour non-renal clearance. There is limited evidence to support the hypothesis that tinzaparin, unlike other LMWHs, does not accumulate in patients with renal insufficiency. 1) Observational studies demonstrated no increase in anti-Xa levels (i.e., no accumulation) when tinzaparin was used for VTE treatment in elderly patients with renal insufficiency. 2) One study showed undetectable LMWH anticoagulant activity by 24 hours after dosing in hemodialysis patients. 3) A systematic review and meta-analysis of the literature in this area performed by our research group found no difference in bleeding and thrombosis complication rates when LMWH (compared to UFH) was used to maintain dialysis circuit patency in patients on hemodialysis.

The current factors which limit the use of tinzaparin in the treatment of patients with VTE and renal insufficiency are: 1) the true risk of accumulation is unknown in a spectrum of patients with varying renal function, and 2) the bleeding risk associated with tinzaparin use is unknown.

Hypothesis. We hypothesize that accumulation during a 5-day course of tinzaparin will not be related to the degree of renal insufficiency.

Study design and methods. We will perform a prospective cohort study of 200 patients with acute VTE, stratified into 4 equal-sized groups by renal function, who will receive initial anticoagulation with tinzaparin for 5 days concurrent with oral anticoagulants. The LMWH anticoagulant effect will be assessed at days 3 and 5 (+/- 1) using trough anti-Xa heparin levels. If accumulation occurs, defined as a trough anti-Xa level > 0.5 IU/mL, the tinzaparin dose will be adjusted according to a nomogram. Patients with an anti-Xa level ≤ 0.5 IU/mL will have no dose adjustment; patients with levels > 0.5 IU/mL will have their tinzaparin dose reduced.

The primary outcome of this study is the proportion of patients in each renal function group with accumulation on or before day 5. We will follow the patients for 48 hours after their final tinzaparin injection. Secondary outcomes are bleeding, recurrent thrombosis, accumulation by day 3, and trough anti-Xa levels > 1.0 IU/mL at any point in the study.

Significance. We hypothesize that tinzaparin does not accumulate in patients with renal insufficiency. However, if accumulation occurs, we hypothesize that dose adjustment according to our novel nomogram will prevent potentially-dangerous levels occurring by day 5. In either case, we will be able to proceed to the next stage in our research plan: an application for funding for a large simple randomized controlled trial examining the safety and efficacy of tinzaparin compared with UFH in patients with renal insufficiency. If accumulation occurs despite the use of the nomogram, then this surrogate outcome suggests that the use of therapeutic-dose tinzaparin is unlikely to be safe in patients with renal insufficiency, a finding which will limit the need to expend further resources on this line of research.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older
* Objectively confirmed VTE requiring anticoagulant therapy, including lower extremity and upper extremity deep vein thrombosis (catheter and non-catheter related, including dialysis access thrombosis [i.e., graft, fistula]); peripheral vein thrombosis (e.g., portal vein, mesenteric vein, cerebral vein thrombosis), and pulmonary embolism

Exclusion Criteria:

* Weight exceeding 105 kg
* Unstable declining renal function, defined as documented change in creatinine > 20% in the past 3 months or clinical circumstances likely to be associated with change in renal function, such as dehydration or severe intercurrent illness. Where no previous creatinine values exist and the patient is otherwise stable, patients will not be excluded on the basis of unknown previous renal function.
* Known allergy to heparin/LMWHs or history of heparin induced thrombocytopenia
* Treatment with UFH, LMWH, danaparoid, oral direct thrombin inhibitors for >48 h
* Bleeding requiring hospitalization or blood transfusion within 6 months(exception is blood transfusion given in relation to surgical procedures within 6 months)
* History of intracerebral hemorrhage
* Known active liver disease (AST or ALT > 3 times the upper limit of normal, or bilirubin > 50 umol/L)
* Known active peptic ulcer disease, with ongoing symptoms or need for anti-ulcer medical therapy
* Thrombocytopenia (platelet count of < 100 x 109/L)
* Ongoing need for antiplatelet agents (clopidogrel, ticlopidine, aspirin > 325 mg daily)
* Pregnancy or lactation
* Geographic inaccessibility
* Unable, or unwilling, to provide written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2005-03; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Anti-Xa level measured on any two of Days 3, 5 or 7 of treatment | Up to 7 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lim, MD, Principal Investigator — St Joseph's Healthcare Hamilton / McMaster University; Mark A Crowther, MD, Principal Investigator — St Joseph's Healthcare Hamilton / McMaster University
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided